CLINICAL TRIAL: NCT00229034
Title: Effect of Activated Protein C and Erythropoietin on the Microvascular Inflammatory Response During Severe Sepsis.
Brief Title: Effect of APC and Epo on the Inflammatory Response During Sepsis
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: R-05-382; 11652E
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Sepsis; Systemic Inflammation
Keywords: Systemic Inflammation; Microvascular Perfusion; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
An observational study to determine the effect of APC and Epo in reducing the systemic inflammatory response during severe sepsis.

DETAILED DESCRIPTION:
An observational study to determine the effect of APC and Epo in reducing the systemic inflammatory response during severe sepsis. Patients already prescribed either drug will be enrolled. The microcirculation of the sublingual vascular bed will be observed with a microscope to detect the alterations in the inflammatory response.

ELIGIBILITY:
Inclusion Criteria:

* patients in the ICU in severe septic shock undergoing APC and/or Epo treatment

Exclusion Criteria:

* any severe comorbid conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the ICU in severe septic shock receiving either APC and/or Epo
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2005-09 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Badhwar, PhD, Principal Investigator — Scientist; Neil Parry, MD, Study Director — Surgeon
Locations (1):
- Lawson Health Research Institute, London, Ontario, Canada